CLINICAL TRIAL: NCT02341339
Title: Utility of Fallopian Tube Cocultures in Assisted Reproductive Technology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WeillMC
Record Dates: First submitted 2014-10-27; First posted 2015-01-19 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fallopian Tube Co-culture (Experimental): fallopian tube biopsy for co-culture of embryos
  Interventions: Procedure: Laparoscopic Surgery (Biopsies of fallopian tube lumen) using a laparoscopic brush/biopsy device

INTERVENTIONS:
Procedure: Laparoscopic Surgery (Biopsies of fallopian tube lumen) using a laparoscopic brush/biopsy device

SUMMARY:
Prospective Feasibility Study:

Fallopian tube cells will be obtained from patients undergoing laparoscopic surgery during their surgical evaluation of infertility. Of note, these patients are already scheduled to undergo surgery as part of their standard of care.

DETAILED DESCRIPTION:
The surgical technique will involve laparoscopic brush and tissue biopsies of the fallopian tube lumen. A small piece of the fallopian tube lining will be removed during the surgery.The biopsy is a minimally invasive and relatively pain free procedure. Co culture blood serum will be drawn at least one day prior to the biopsy and during the IVF cycle. The fallopian tube sample is sent to the Center for Reproductive Medicine (CRM) lab where it is treated, purified and frozen. The next month or whenever the physician deems appropriate, the patient will then undergo a typical IVF cycle and will be given standard medication protocol determined by her physician to stimulate egg growth in her ovaries. The patient's eggs will be retrieved and mixed with sperm. At this time, the lab will begin to thaw and grow the fallopian tube cells. Once fertilization is confirmed, the patient's embryos will be placed on top of her own (now thawed) fallopian tube cells and allowed to grow. Subsequently, the embryos will be placed on top of her uterus for implantation and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing assisted reproductive technology at Weill Cornell Medical College (WCMC) and are scheduled to undergo surgery as part of their standard of care
* Women who had a prior failed IVF cycle
* Women with normal Hysterosalpingogram (HSG) or a prior laparoscopy confirming normal tubal status
* Both the patient (potential subject) and her partner must sign the consent form

Exclusion Criteria:

* Pregnancy
* Undiagnosed vaginal bleeding
* Fallopian tube disease

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with good embryo quality as a measure of efficacy | 8 weeks
  The outcomes measures for embryo quality will include an assessment of the embryo grade, embryo fragmentation rates, implantation rates and pregnancy rates.

SECONDARY OUTCOMES:
Number of participants with Adverse Events as a measure of Safety and Tolerability | 8 weeks
  We will assess the incidence of pain, bleeding and infection rates

CONTACTS AND LOCATIONS:
Overall Officials: Rony Elias, MD, Principal Investigator — Weill Medical College of Cornell University